CLINICAL TRIAL: NCT00791024
Title: Phase One Study and Two of a New Method for Local Analgesia
Brief Title: Development of a New Method for Analgesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ove Andersen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, Research director, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRC06
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Analgesia
Keywords: Analgesia Tests; Analog Pain Scale; Pain Measurement
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: CRC-Pharma 001; Drug: lidocaine suspension

INTERVENTIONS:
Drug: CRC-Pharma 001 — 50 mg
Drug: lidocaine suspension — 5.0 ml lidocaine suspension(20mg/ml) adm. 10 min. before oesophagogastroduodenoscopy.

SUMMARY:
Aim: To examine a new method to perform local anesthesia in order to diminish the inconvenience by the procedure in patients before performing intubation or oesophagogastroduodenoscopy.

DETAILED DESCRIPTION:
A phase one and two study. part one is performed as a single arm unblinded uncontrolled study in 16 obese patients undergoing awake intubation (investigational pill). The second part is a phase two study randomized single blinded study in 100 patient attending a day case endoscopy unit for oesophagogastroduodenoscopy (investigational pill versus lidocaine suspension).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for adipositas surgery
* Patients who attend for oesophagogastroduodenoscopy.

Exclusion Criteria:

* Severe psychiatric diseases
* Alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
VAS score | at day O and 3

SECONDARY OUTCOMES:
Questionnaire( examiner and patient) | performed at day 0 and 3

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University, Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Mogensen S, Pulis S, Kristensen BB, Ravn L, Treldal C, Rasmussen M, Mogensen T, Andersen O. A new method to facilitate oro-tracheal intubation of awake patients: a pilot study. Eur J Anaesthesiol. 2012 Nov;29(11):546-7. doi: 10.1097/EJA.0b013e328357e4e5. No abstract available. PMID 22955296